CLINICAL TRIAL: NCT06951750
Title: Effect of Foot Reflexology on Postpartum Afterpains
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hala Ismail Mahmoud, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005673
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Pain, Labor
MeSH Terms: conditions — Labor Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reflexology group (Experimental): The participants will receive reflexology on foot and on specific uterine points in the first hour post-partum and will be repeated in the second hour post-partum
  Interventions: Other: Reflexology; Other: general foot massage
- Placebo reflexology (Active Comparator): The participants will receive reflexology on foot and on heel (placebo points) in the first hour post-partum and will be repeated in the second hour post-partum
  Interventions: Other: placebo reflexology; Other: general foot massage

INTERVENTIONS:
Other: Reflexology — The participants will receive two minutes of specific reflexology on each point of the uterus, pituitary, and solar plexus in the form of rotational pressures. This will be performed in the first hour post-partum and will be repeated in the second hour post-partum
  Arms: Reflexology group
Other: placebo reflexology — The participants will receive rotational pressures on a neutral point on the lateral side of the heel (placebo point) for six minutes. This will be performed in the first hour post-partum and will be repeated in the second hour post-partum
  Arms: Placebo reflexology
Other: general foot massage — The participants will receive a general massage on each foot for four minutes. This will be performed in the first hour post-partum and will be repeated in the second hour post-partum

SUMMARY:
This study will be conducted to determine the effect of foot reflexology on afterpains after normal labor.

DETAILED DESCRIPTION:
Afterpains are among the most prevalent complaints after natural vaginal delivery. Non-pharmacological treatment modalities to relieve afterpains are an important care priority as they can lead to maternal and neonatal complications including anxiety, sleep disturbances, emotional disorders, depression, inability to care for the baby and continue breastfeeding, delays in early breastfeeding, reduced maternal ability to perform daily chores.

It was reported that pain in the early hours postpartum is one of the most important factors contributing to chronic postpartum pain and depression. Furthermore, pain and stress increase adrenaline release and decrease oxytocin release, thus leading to the cessation of the oxytocin reflex and disrupting breast milk production in addition to causing discomfort for the mother.

Since afterpains is a common problem that affects the physical and mental well-being of mothers, it requires the attention of healthcare providers. There is only one study that investigated the effect of reflexology on the pain level of afterpains after normal vaginal delivery. Moreover, no study investigated the effect of reflexology on either the behavioral response toward pain or the pressure pain threshold. Therefore, this study will be conducted to provide physiotherapists with updated scientific Knowledge concerning the effect of foot reflexology on afterpains after normal labor. This Study may expand the role of physiotherapy in women's health.

ELIGIBILITY:
Inclusion Criteria:

* They will be multipara (2-3).
* They will be normal vaginal labor

Exclusion Criteria:

* High-risk pregnancy.
* Post-partum hemorrhage.
* Neonatal birth weight over 4 kg.
* Over distension of the uterus.
* Cesarean section.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of pain intensity | 4 hours
  It will be used to assess pain levels in women in both groups before treatment (1 hour postpartum), after 2 hours, 3 hours and 4 hours postpartum. It comprises 16 items that reflect equally the sensory (11 items) and affective (5 items) dimensions of pain. These items were responded to by 5 points Likert-like scale as follows: 0 = none, 1= Mild, 2 = Moderate 3 =Severe, 4 = Unbearable pain. The total score will be ranged between 0 to 60 and classified as follows: No pain = 0, mild pain (from 1 to 15), moderate pain (from 16 to 30), severe pain (from 31 to 45), and unbearable pain (from 46 to 60). These pain-rating scales have shown good validity and reliability for assessing pain intensity. The intraclass correlation coefficients were 0.95
Modified version of chamber price pain Rating Scale | 4 hours
  This tool was adapted for measuring any behavioral responses towards pain including 4 dimensions: Gross motor activity, posture, verbalization, and facial expression. For each dimension, one of 3 alternatives (0, 1, and 2) is to be elicited by the researcher. For posture, the alternatives are very relaxed, guarded, and tense posture. For gross motor activity, the alternatives are very restless, slightly restless, and quiet. For facial expression, alternatives are not frowning, some frowning, and constant frowning or grimacing. Lastly, women's verbalization differs between normal, no sound, groans/moans, and cries/sobs. The total score of the 4 dimensions varies between 0-8 and is categorized as follows: no pain (0) mild pain (1-2), moderate pain (3-4), severe pain (5-6), and intolerable pain (7- 8). it will be measured for both groups before treatment (1 hour postpartum), after 2 hours, 3 hours and 4 hours postpartum.
Pressure pain threshold (PPT): | 4 hours
  The pressure algometer will be used to measure deep muscular tissue sensitivity for participants in both groups before treatment (1 hour postpartum), after 2 hours, 3 hours and 4 hours postpartum.. The test determines the amount of pressure over a given area in which a steadily increasing no-painful-pressure stimulus turns into a painful pressure sensation. A varying pressure is applied from 0.5 to 1 kg/sec in a perpendicular direction relative to the muscle. Six points will be determined to evaluate the PPTs. PPT recording sites will be marked out the abdomen around the umbilical scar and lumbar region as follows: Two measurements 4 cm from the umbilicus, bilaterally (points I and II), two other measurements 4 cm below the previous ones (points III and IV), a single measurement 4 cm from the lower margin of the umbilicus (point V) and another single measurement into the medial side of the lumbar region below the fifth lumbar vertebra, correspond-in to S2-S4 (point VI).

CONTACTS AND LOCATIONS:
Overall Officials: Hazem El-Ashmawy, Professor, Study Director — Cairo University; Doaa Osman, As professor, Study Chair — Cairo University
Locations (1):
- Hala Ismail Mahmoud, Cairo, Egypt